CLINICAL TRIAL: NCT00778934
Title: A Single-blind, Multi-center, In-home Use Study to Evaluate Sexual Enhancement Effects of Product PD-F-5394 in Females
Brief Title: In-Home Use Study to Evaluate Use of an Intimate Health Product in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: CA-P-5739-1
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Coitus
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Intimate Health Gel
  Interventions: Other: Intimate Health Gel

INTERVENTIONS:
Other: Intimate Health Gel — Intimate Health Gel
  Other Names: Not marketed yet

SUMMARY:
The purpose of this study is to evaluate the effects of an intimate health product on sexual experience in females.

DETAILED DESCRIPTION:
Study to evaluate consumer perceptions of a cosmetic intimate health product on sexual experience in females, using a validated psychometric questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy females >18 years of age
* In committed heterosexual relationship for >6months
* Of adequate sexual functioning
* On acceptable method of birth control

Exclusion Criteria:

* Pregnant or breastfeeding
* Allergy to product ingredients
* Irritation or infection in genital area
* Unstable or uncontrolled medical condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To assess the effect of product on sexual enhancement by comparing baseline questionnaire responses to the end of study questionnaire responses | End of study (3 weeks after baseline visit)

SECONDARY OUTCOMES:
Safety Assessments will consist of monitoring and recording all non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs), their frequency, severity, seriousness, and relationship to the investigational product. | throughout duration of the study (+ 30 days for spontaneously reported SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Wanser, Study Director — J&J CPPW
Locations (2):
- United States (2):
  - Center of Marital and Sexual Health of South Florida, West Palm Beach, Florida
  - Center for Marital and Sexual Health, Inc., Beachwood, Ohio